CLINICAL TRIAL: NCT03568110
Title: The Impact of Frailty on the Postoperative Outcomes of Gastric Cancer Surgery
Brief Title: Frailty and Postoperative Outcomes After Gastric Cancer Surgery
Acronym: TOREGA
Status: Completed | Type: Observational
Sponsor: Parc de Salut Mar (Other)
Responsible Party: Principal Investigator, Manuel Ramón Pera Román, Professor of Surgery, Head of Section of Gastrointestinal Surgery, Parc de Salut Mar
Other Study IDs: 1
Record Dates: First submitted 2018-05-09; First posted 2018-06-26 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Gastric Cancer; Frail Elderly Syndrome; Postoperative Complications; Quality of Life
MeSH Terms: conditions — Stomach Neoplasms; Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Background. Gastric cancer is an important health care problem even though treatment advances, and it is diagnosed mainly in elderly. Surgery is the main treatment for gastric cancer and is associated with a high rate of postoperative complications and mortality, even higher in older patients. Chronological age seems not to be the main factor influencing the worse outcome of older patients, comorbidities and frailty have also been taken into account recently.

Methods. Participation in the study will be offered to all centers that are currently part of the Spanish EURECCA (EUropean REgistry of Cancer CAre) Esophagogastric Cancer Registry. The impact of the frailty on different outcome variables will be evaluated. The main outcome variable will be 90-day mortality after the intervention. Health-Related Quality of Life (HRQoL) will also be evaluated.

Objective. The objective of the study is to value the impact of frailty on gastric cancer surgery outcomes therein the Spanish EURECCA Esophagogastric Cancer Registry.

DETAILED DESCRIPTION:
Introduction

Gastric cancer is the fifth most frequent cancer and the third cause of death due to cancer. The increase in life expectancy cause it to be diagnosed more and more in elderly people, with an average age at diagnosis of 68 years in the West.

Surgery is the main treatment for gastric cancer and is associated with a high rate of postoperative complications and mortality, which is even higher in elderly patients (data from the ACS-NSQIP between 2007 and 2013: 30-day severe morbidity from 16.3% in 80 years and 30-day mortality from 1.2% in 80 years).

Generally, advanced chronological age is considered a negative prognostic factor for complications and hospital stay in major surgery. Age per se, however, seems to be responsible only in part for the increased risk of postoperative complications.

Greater risks seem to be associated with other factors such as comorbidities, so, in the preoperative evaluation, variables such as the Charlson comorbidity index have been introduced. Another variable that has emerged recently for the estimation of perioperative risk is frailty, which is defined as "a medical syndrome with multiple causes and contributors that is characterized by a decrease in strength, endurance and physiological capacity, which increases the risk of the vulnerability of the individual and/or death". Surgery is a major stress factor that can disrupt physiological homeostasis; therefore, frailty has a clinical significance when considering surgery in elderly patients.

There are two main ways to measure frailty: one by clinical definitions of a fragile phenotype and another by frailty indexes that assess the accumulated deficits in multiple domains. Measures to assess frailty are numerous and this is a limitation when standardizing and comparing studies; among the most used there are the Fried criteria, the frailty index of the Canadian Study of Health and Aging (CSHA-FI) and the modified frailty index of Velanovich (mFI: modified Frailty Index).

Other indices widely used in the clinic are the Geriatric 8 (G8), which is recommended above all in elderly patients with cancer and the Groningen index (GFI: Groningen Frailty Indicator). The prevalence of frailty in elderly patients (65 years or older) is highly variable, probably due to the diversity in the definitions of frailty (4.0-59.1% in community residences, 10.4-56.0% in patients who are candidates for elective surgery) (18, 19, 20). The prevalence of frailty increases in females and with age (being 15.7% in patients aged 80-84 years and 26.1% in patients older than 85 years).

Frailty appears in several studies as a more important indicator than chronological age with respect to postoperative results. There are evidences that relate frailty, evaluated with different indices, with the increase of postoperative complications, hospital stay, need of discharge to convalescence centers, health costs, short and long term mortality, after major surgery.

Therefore, it is important to identify fragile patients to implement prevention programs through global geriatric assessments (CGA Comprehensive Geriatric Assessment). Just by having more clinical attention for more fragile patients after major surgery there can be better results of short and long-term postoperative mortality. Likewise, as demonstrated in randomized clinical studies, prehabilitation and global geriatric assessment programs improve the results in terms of postoperative complications and hospital stay.

The CGA is an established method to evaluate and optimize the physical state, the psychological, functional and social problems in elderly patients in order to improve the results of the treatments. It implies an interdisciplinary evaluation of multiple domains, followed by planning for analysis, treatment, rehabilitation and long-term follow-up.

This allows, in the first place, to intervene before an operation, to increase the physiological reserve of a patient, especially with exercise and nutrition. In addition, the therapeutic decision can be guided by adapting the surgical recommendations to the physiological capacity of the patient; second, the knowledge of the increased risk of complications and the possible need for transfer to institutions (especially in patients who live alone) prepares patients and their families for postoperative evolution.

The majority of studies published in the literature on the relationship between frailty and postoperative results are retrospective studies, which evaluate populations of patients undergoing major surgery and who, in general, analyze short-term results (30-day mortality). None of these takes into account the impact of surgery on the quality of life of this group of patients. Among all these studies there is very little information about the influence of frailty in gastric cancer surgery. There is only one retrospective study that focuses only on gastric cancer surgery, using the Groningen index and revealing an increase in in-hospital mortality and serious complications (Clavien-Dindo complications score ≥ 3) in fragile patients.

Objective

The aim of the present study is to assess the impact of frailty on the results of gastric cancer surgery (long-term postoperative morbidity and mortality, hospital stay, readmissions, need of transfer to institution of medium or long stay and quality of life).

Methods

This is a prospective and multicenter cohort study, within the Spanish EURECCA Esophagogastric Cancer Project, to investigate the impact of frailty on the postoperative results of surgery for gastric cancer in elderly patients.

Participation in the study will be offered to all centers that are currently part of the Spanish EURECCA Esophagogastric Cancer Registry. Those hospitals that show their desire to participate must sign the Letter of Commitment.

The impact of the frailty on different outcome variables will be evaluated. The main outcome variable will be 90-day mortality after the intervention. Other secondary outcome variables will also be evaluated: incidence of serious complications (Clavien-Dindo complications score ≥ 3), Complication Comprehensive Index (CCI) score, hospital stay, incidence of death in patients suffering from a complication (failure-to-rescue), hospital readmission within the first 30 days after the discharge, destination of the patient after discharge from hospital [home, social health centers, or geriatric residence], mortality at 12 months after the intervention, quality of life before the intervention and at 12 months.

For the assessment of frailty (frailty screening), two questionnaires will be used:

* Questionnaire G8: This is a questionnaire with 8 questions, easy to use, with a total score that varies from 0 to 17 points. Previous studies suggest the score ≤ 14 as a cut-off point to identify the fragile patient, with a sensitivity of 92% and specificity of 52%.
* Modified frailty index: This index was described by Velanovich et al., based on a previously validated simplification of the frailty index CSHAFI (Canadian Study of Health and Aging Frailty Index), which was specifically designed to analyze data included in the National Surgical Quality Improvement Program of the American College of Surgeons (ACSNSQIP). It consists of 11 questions with 1 point assigned to each of them on the functional, endocrine, respiratory, cardiovascular and neurological status of the patient. It allows to divide the patients into 4 groups: without frailty (FI = 0), slightly fragile (FI = 1), moderately fragile (FI = 2) and severely fragile (FI ≥ 3).

Postoperative complications will be classified according to the recommendations proposed by the European Chapter of the International Gastric Cancer Association (EGCA) (unpublished data), its severity through the classification of Clavien-Dindo and the CCI. In particular, the CCI will be calculated using the free application that can be found on the website: www.assessurgery.com/calculator_single/.

Health-Related Quality of Life (HRQoL) will be evaluated with the validated Quality of Life questionnaires of the European Organization for Research and Treatment of Cancer (EORTC-QLQ), QLQ-C30 (30 items Core Quality of Life Questionnaire, version 3.0) and with the specific module for gastric cancer QLQ-STO22 (22 items Stomach Quality of Life Questionnaire). The permission for its use by the EORTC is available.

* The EORTC-QLQ-C30 is a questionnaire that reflects the multidimensionality of HRQoL in patients with cancer. It is composed of 30 questions distributed in five functional scales (physical, role, cognitive, emotional and social), three scales of symptoms (fatigue, pain and nausea and vomiting), a global health scale and a series of additional questions to evaluate symptoms commonly referred by patients diagnosed with cancer (dyspnea, loss of appetite, insomnia, constipation and diarrhea) and the perceived financial impact.
* The EORTC-QLQ-STO22 questionnaire contains 22 structured items in five domains (dysphagia, food restrictions, pain, reflux and anxiety) and four specific items (dry mouth, alteration of taste perception, body image and hair loss) related to the symptoms of the disease.

The calculation of the sample size is based on the primary objective of comparing fragile versus non-fragile patients with respect to postoperative mortality at 90 days after the intervention. Based on mortality data previously published in a retrospective study by Mosquera et al., it is estimated that mortality for the group of non-frail patients is 0.6% and for the group with frailty 4.3%. From the data of the literature, a prevalence of 23% of frailty is calculated in the population of patients with gastric cancer and age ≥ 70 years undergoing gastrectomy.

For a power of 80% and a level of significance of 95% in a unilateral analysis, it is estimated that 276 non-fragile patients and 92 fragile patients would be needed to detect as statistically significant the difference between the proportion of patients who die between both groups.

The characteristics of fragile and non-fragile patient groups will be compared through frequency tables. The Chi-square test will be used to compare the differences between the categorical variables and the ANOVA test for the continuous variables. Different analyzes are proposed according to the study variables that are to be analyzed. For dichotomous type response variables (90- day mortality, 12-month mortality, incidence of serious complications, incidence of in-hospital death in patients with complications, and hospital readmission at 30 days after discharge), a multivariate logistic regression will be used to evaluate the risk (odds ratio) of these variables. For continuous response variables (ICC score) at 30 days after the intervention, and number of days of hospital stay), linear regression models will be used. For the variable categorical response of the patient after hospital discharge, an ordinal logistic regression model will be done. All regression models will be adjusted for age, sex, body mass index (BMI), type of gastrectomy, center volume, neoadjuvant treatment and degree of frailty. Regarding HRQoL analysis, the mean scores and 95% confidence intervals for the different domains of preoperative HRQoL and one year after surgery will be calculated. Changes of more than 10 points on a scale from 0 to 100 will be considered clinically relevant as previously suggested in other publications.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 70 years patients diagnosed with gastric cancer candidates for radical resection

Exclusion Criteria:

* metastatic patients
* patients candidates for palliative treatment
* patients without a signed informed consent

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: The possibility to participate to the study will be offered to all the hospitals members of the Spanish EURECCA Esophagogastric Cancer Registry. The hospitals that will participate must sign a commitment. Every patient that fit the eligibility criteria will be part of the study.
Sampling Method: Non-Probability Sample
Enrollment: 432 (Actual)
Dates: Start 2019-03-05 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
90-day mortality | 90 days after surgery
  Mortality at 90 days after surgery

SECONDARY OUTCOMES:
Severe complications | 30 days after surgery
  Postoperative complications Clavien-Dindo score ≥ III
  Clavien-Dindo score:
  Grade I Any deviation from the normal postoperative course without the need for pharmacological treatment or surgical, endoscopic and radiological interventions
  Grade II Requiring pharmacological treatment with drugs other than such allowed for grade I complications
  Grade III Requiring surgical, endoscopic or radiological intervention
  * IIIa Intervention not under general anesthesia
  * IIIb Intervention under general anesthesia
  Grade IV Life-threatening complication requiring Intensive Care Unit-management
  * IVa single organ dysfunction (including dialysis)
  * IVb multiorgandysfunction Grade V Death of a patient
  Higher values represent a worse outcome.
Complication Comprehensive Index | 30 days after surgery
  Complication Comprehensive Index from www.assessurgery.com/calculator_single/
  The CCI® calculator is an online tool to support the assessment of patients' overall morbidity. The Comprehensive Complication Index (CCI®) is based on the complication grading by Clavien-Dindo Classification and implements every occurred complication after an intervention. The overall morbidity is reflected on a scale from 0 (no complication) to 100 (death). CCI® =√ (wC1 + wC2 ...+ wCx ) /2.
  Higher values represent a worse outcome.
Failure to rescue | 30 days after surgery
  Postoperative death after a treatable complication
Hospital stay | 30 days after surgery
  Number of days of hospital stay
Patient discharge facility | 30 days after surgery
  Facility where the patient goes after the hospital stay
Readmission | 30 days after discharge
  Readmission within 30 days after discharge
12-month mortality | 12 months after surgery
  Mortality at 12 months after surgery
Health-related Quality of life before the intervention (EORTC-QLQ-C30) | 2 weeks before surgery
  Quality of life before the intervention evaluated with the EORTC (European Organization for Research and Treatment of Cancer) QLQ-C30 questionnaire:
  - The EORTC-QLQ-C30 (30 items Core Quality of Life Questionnaire) includes five functional scales, three symptom scales, a global health status/QoL scale, and six single items. All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level (a high/healthy level of functioning in functional scales, a high Quality of Life in Quality of Life scales, a high level of symptomatology/problems in symptom scales).
Health-related Quality of life before the intervention (EORTC-QLQ-STO22) | 2 weeks before surgery
  Quality of life before the intervention evaluated with the EORTC (European Organization for Research and Treatment of Cancer) QLQ-STO22 questionnaire:
  - The QLQ-STO22 (22 items Stomach Quality of Life Questionnaire) consists of five multi-item symptoms scales and four single symptoms items. All of the scales and single-item measures range in score from 0 to 100. Higher scores represent greater level of symptoms.
Health-related Quality of life at 12 months (EORTC-QLQ-C30) | 12 months after surgery
  Quality of life before the intervention evaluated with the EORTC (European Organization for Research and Treatment of Cancer) QLQ-C30 questionnaire:
  - The EORTC-QLQ-C30 (30 items Core Quality of Life Questionnaire) includes five functional scales, three symptom scales, a global health status/QoL scale, and six single items. All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level (a high/healthy level of functioning in functional scales, a high Quality of Life in Quality of Life scales, a high level of symptomatology/problems in symptom scales).
Health-related Quality of life at 12 months (EORTC-QLQ-STO22) | 12 months after surgery
  Quality of life before the intervention evaluated with the EORTC (European Organization for Research and Treatment of Cancer) QLQ-STO22 questionnaire:
  - The QLQ-STO22 (22 items Stomach Quality of Life Questionnaire) consists of five multi-item symptoms scales and four single symptoms items. All of the scales and single-item measures range in score from 0 to 100. Higher scores represent greater level of symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Manuel Pera, Principal Investigator — Parc de Salut Mar
Locations (1):
- H. U. Germans Trias i Pujol, Badalona, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hamilton TD, Mahar AL, Haas B, Beyfuss K, Law CHL, Karanicolas PJ, Coburn NG, Hallet J. The impact of advanced age on short-term outcomes following gastric cancer resection: an ACS-NSQIP analysis. Gastric Cancer. 2018 Jul;21(4):710-719. doi: 10.1007/s10120-017-0786-6. Epub 2017 Dec 11. PMID 29230588
- [Background] Polanczyk CA, Marcantonio E, Goldman L, Rohde LE, Orav J, Mangione CM, Lee TH. Impact of age on perioperative complications and length of stay in patients undergoing noncardiac surgery. Ann Intern Med. 2001 Apr 17;134(8):637-43. doi: 10.7326/0003-4819-134-8-200104170-00008. PMID 11304103
- [Background] Kim SW, Han HS, Jung HW, Kim KI, Hwang DW, Kang SB, Kim CH. Multidimensional frailty score for the prediction of postoperative mortality risk. JAMA Surg. 2014 Jul;149(7):633-40. doi: 10.1001/jamasurg.2014.241. PMID 24804971
- [Background] Tegels JJ, Stoot JH. Way forward: Geriatric frailty assessment as risk predictor in gastric cancer surgery. World J Gastrointest Surg. 2015 Oct 27;7(10):223-5. doi: 10.4240/wjgs.v7.i10.223. PMID 26523209
- [Background] Partridge JS, Harari D, Dhesi JK. Frailty in the older surgical patient: a review. Age Ageing. 2012 Mar;41(2):142-7. doi: 10.1093/ageing/afr182. PMID 22345294
- [Background] Morley JE, Vellas B, van Kan GA, Anker SD, Bauer JM, Bernabei R, Cesari M, Chumlea WC, Doehner W, Evans J, Fried LP, Guralnik JM, Katz PR, Malmstrom TK, McCarter RJ, Gutierrez Robledo LM, Rockwood K, von Haehling S, Vandewoude MF, Walston J. Frailty consensus: a call to action. J Am Med Dir Assoc. 2013 Jun;14(6):392-7. doi: 10.1016/j.jamda.2013.03.022. PMID 23764209
- [Background] Fried LP, Tangen CM, Walston J, Newman AB, Hirsch C, Gottdiener J, Seeman T, Tracy R, Kop WJ, Burke G, McBurnie MA; Cardiovascular Health Study Collaborative Research Group. Frailty in older adults: evidence for a phenotype. J Gerontol A Biol Sci Med Sci. 2001 Mar;56(3):M146-56. doi: 10.1093/gerona/56.3.m146. PMID 11253156
- [Background] Rockwood K, Mitnitski A. Frailty in relation to the accumulation of deficits. J Gerontol A Biol Sci Med Sci. 2007 Jul;62(7):722-7. doi: 10.1093/gerona/62.7.722. PMID 17634318
- [Background] McIsaac DI, Bryson GL, van Walraven C. Association of Frailty and 1-Year Postoperative Mortality Following Major Elective Noncardiac Surgery: A Population-Based Cohort Study. JAMA Surg. 2016 Jun 1;151(6):538-45. doi: 10.1001/jamasurg.2015.5085. PMID 26791334
- [Background] Rockwood K, Song X, MacKnight C, Bergman H, Hogan DB, McDowell I, Mitnitski A. A global clinical measure of fitness and frailty in elderly people. CMAJ. 2005 Aug 30;173(5):489-95. doi: 10.1503/cmaj.050051. PMID 16129869
- [Background] Velanovich V, Antoine H, Swartz A, Peters D, Rubinfeld I. Accumulating deficits model of frailty and postoperative mortality and morbidity: its application to a national database. J Surg Res. 2013 Jul;183(1):104-10. doi: 10.1016/j.jss.2013.01.021. Epub 2013 Feb 1. PMID 23415494
- [Background] Bellera CA, Rainfray M, Mathoulin-Pelissier S, Mertens C, Delva F, Fonck M, Soubeyran PL. Screening older cancer patients: first evaluation of the G-8 geriatric screening tool. Ann Oncol. 2012 Aug;23(8):2166-2172. doi: 10.1093/annonc/mdr587. Epub 2012 Jan 16. PMID 22250183
- [Background] Smets IH, Kempen GI, Janssen-Heijnen ML, Deckx L, Buntinx FJ, van den Akker M. Four screening instruments for frailty in older patients with and without cancer: a diagnostic study. BMC Geriatr. 2014 Feb 26;14:26. doi: 10.1186/1471-2318-14-26. PMID 24571290
- [Background] Collard RM, Boter H, Schoevers RA, Oude Voshaar RC. Prevalence of frailty in community-dwelling older persons: a systematic review. J Am Geriatr Soc. 2012 Aug;60(8):1487-92. doi: 10.1111/j.1532-5415.2012.04054.x. Epub 2012 Aug 6. PMID 22881367
- [Background] Robinson TN, Wu DS, Pointer L, Dunn CL, Cleveland JC Jr, Moss M. Simple frailty score predicts postoperative complications across surgical specialties. Am J Surg. 2013 Oct;206(4):544-50. doi: 10.1016/j.amjsurg.2013.03.012. Epub 2013 Jul 20. PMID 23880071
- [Background] Makary MA, Segev DL, Pronovost PJ, Syin D, Bandeen-Roche K, Patel P, Takenaga R, Devgan L, Holzmueller CG, Tian J, Fried LP. Frailty as a predictor of surgical outcomes in older patients. J Am Coll Surg. 2010 Jun;210(6):901-8. doi: 10.1016/j.jamcollsurg.2010.01.028. Epub 2010 Apr 28. PMID 20510798
- [Background] Robinson TN, Wallace JI, Wu DS, Wiktor A, Pointer LF, Pfister SM, Sharp TJ, Buckley MJ, Moss M. Accumulated frailty characteristics predict postoperative discharge institutionalization in the geriatric patient. J Am Coll Surg. 2011 Jul;213(1):37-42; discussion 42-4. doi: 10.1016/j.jamcollsurg.2011.01.056. Epub 2011 Mar 23. PMID 21435921
- [Background] Hall DE, Arya S, Schmid KK, Carlson MA, Lavedan P, Bailey TL, Purviance G, Bockman T, Lynch TG, Johanning JM. Association of a Frailty Screening Initiative With Postoperative Survival at 30, 180, and 365 Days. JAMA Surg. 2017 Mar 1;152(3):233-240. doi: 10.1001/jamasurg.2016.4219. PMID 27902826
- [Background] Fagard K, Leonard S, Deschodt M, Devriendt E, Wolthuis A, Prenen H, Flamaing J, Milisen K, Wildiers H, Kenis C. The impact of frailty on postoperative outcomes in individuals aged 65 and over undergoing elective surgery for colorectal cancer: A systematic review. J Geriatr Oncol. 2016 Nov;7(6):479-491. doi: 10.1016/j.jgo.2016.06.001. Epub 2016 Jun 21. PMID 27338516
- [Background] Mosquera C, Spaniolas K, Fitzgerald TL. Impact of frailty on surgical outcomes: The right patient for the right procedure. Surgery. 2016 Aug;160(2):272-80. doi: 10.1016/j.surg.2016.04.030. Epub 2016 Jun 3. PMID 27267548
- [Background] Tegels JJ, de Maat MF, Hulsewe KW, Hoofwijk AG, Stoot JH. Value of geriatric frailty and nutritional status assessment in predicting postoperative mortality in gastric cancer surgery. J Gastrointest Surg. 2014 Mar;18(3):439-45; discussion 445-6. doi: 10.1007/s11605-013-2443-7. Epub 2014 Jan 14. PMID 24420730
- [Background] Augustin T, Burstein MD, Schneider EB, Morris-Stiff G, Wey J, Chalikonda S, Walsh RM. Frailty predicts risk of life-threatening complications and mortality after pancreatic resections. Surgery. 2016 Oct;160(4):987-996. doi: 10.1016/j.surg.2016.07.010. Epub 2016 Aug 18. PMID 27545992
- [Background] Vermillion SA, Hsu FC, Dorrell RD, Shen P, Clark CJ. Modified frailty index predicts postoperative outcomes in older gastrointestinal cancer patients. J Surg Oncol. 2017 Jun;115(8):997-1003. doi: 10.1002/jso.24617. Epub 2017 Apr 24. PMID 28437582
- [Background] Hewitt J, Moug SJ, Middleton M, Chakrabarti M, Stechman MJ, McCarthy K; Older Persons Surgical Outcomes Collaboration. Prevalence of frailty and its association with mortality in general surgery. Am J Surg. 2015 Feb;209(2):254-9. doi: 10.1016/j.amjsurg.2014.05.022. Epub 2014 Jul 27. PMID 25173599
- [Background] Obeid NM, Azuh O, Reddy S, Webb S, Reickert C, Velanovich V, Horst HM, Rubinfeld I. Predictors of critical care-related complications in colectomy patients using the National Surgical Quality Improvement Program: exploring frailty and aggressive laparoscopic approaches. J Trauma Acute Care Surg. 2012 Apr;72(4):878-83. doi: 10.1097/TA.0b013e31824d0f70. PMID 22491599
- [Background] Abdullah HR, Lien VP, Ong HK, Er PL, Hao Y, Khan SA, Liu CW. Protocol for a single-centre, randomised controlled study of a preoperative rehabilitation bundle in the frail and elderly undergoing abdominal surgery. BMJ Open. 2017 Aug 4;7(8):e016815. doi: 10.1136/bmjopen-2017-016815. PMID 28778994
- [Background] Huddleston JM, Long KH, Naessens JM, Vanness D, Larson D, Trousdale R, Plevak M, Cabanela M, Ilstrup D, Wachter RM; Hospitalist-Orthopedic Team Trial Investigators. Medical and surgical comanagement after elective hip and knee arthroplasty: a randomized, controlled trial. Ann Intern Med. 2004 Jul 6;141(1):28-38. doi: 10.7326/0003-4819-141-1-200407060-00012. PMID 15238368
- [Background] Macpherson DS, Lofgren RP. Outpatient internal medicine preoperative evaluation: a randomized clinical trial. Med Care. 1994 May;32(5):498-507. doi: 10.1097/00005650-199405000-00008. PMID 8182977
- [Background] Partridge JS, Harari D, Martin FC, Dhesi JK. The impact of pre-operative comprehensive geriatric assessment on postoperative outcomes in older patients undergoing scheduled surgery: a systematic review. Anaesthesia. 2014 Jan;69 Suppl 1:8-16. doi: 10.1111/anae.12494. PMID 24303856
- [Background] Li C, Carli F, Lee L, Charlebois P, Stein B, Liberman AS, Kaneva P, Augustin B, Wongyingsinn M, Gamsa A, Kim DJ, Vassiliou MC, Feldman LS. Impact of a trimodal prehabilitation program on functional recovery after colorectal cancer surgery: a pilot study. Surg Endosc. 2013 Apr;27(4):1072-82. doi: 10.1007/s00464-012-2560-5. Epub 2012 Oct 9. PMID 23052535
- [Background] Hulzebos EH, Smit Y, Helders PP, van Meeteren NL. Preoperative physical therapy for elective cardiac surgery patients. Cochrane Database Syst Rev. 2012 Nov 14;11(11):CD010118. doi: 10.1002/14651858.CD010118.pub2. PMID 23152283
- [Background] Baitar A, Van Fraeyenhove F, Vandebroek A, De Droogh E, Galdermans D, Mebis J, Schrijvers D. Evaluation of the Groningen Frailty Indicator and the G8 questionnaire as screening tools for frailty in older patients with cancer. J Geriatr Oncol. 2013 Jan;4(1):32-8. doi: 10.1016/j.jgo.2012.08.001. Epub 2012 Aug 24. PMID 24071490
- [Background] Dindo D, Demartines N, Clavien PA. Classification of surgical complications: a new proposal with evaluation in a cohort of 6336 patients and results of a survey. Ann Surg. 2004 Aug;240(2):205-13. doi: 10.1097/01.sla.0000133083.54934.ae. PMID 15273542
- [Background] Slankamenac K, Nederlof N, Pessaux P, de Jonge J, Wijnhoven BP, Breitenstein S, Oberkofler CE, Graf R, Puhan MA, Clavien PA. The comprehensive complication index: a novel and more sensitive endpoint for assessing outcome and reducing sample size in randomized controlled trials. Ann Surg. 2014 Nov;260(5):757-62; discussion 762-3. doi: 10.1097/SLA.0000000000000948. PMID 25379846
- [Background] Schwarz R, Hinz A. Reference data for the quality of life questionnaire EORTC QLQ-C30 in the general German population. Eur J Cancer. 2001 Jul;37(11):1345-51. doi: 10.1016/s0959-8049(00)00447-0. PMID 11435063
- [Background] Avery K, Hughes R, McNair A, Alderson D, Barham P, Blazeby J. Health-related quality of life and survival in the 2 years after surgery for gastric cancer. Eur J Surg Oncol. 2010 Feb;36(2):148-54. doi: 10.1016/j.ejso.2009.09.008. PMID 19836921

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-16): https://cdn.clinicaltrials.gov/large-docs/10/NCT03568110/Prot_SAP_000.pdf